CLINICAL TRIAL: NCT05831605
Title: Success Rate Comparison of Venipuncture in Children With and Without Near-infrared Light
Acronym: ALPIVEINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D20170121; ID-RCB (Registry Identifier: 2022-A02584-39)
Record Dates: First submitted 2023-03-27; First posted 2023-04-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-06

CONDITIONS: Venipuncture
Keywords: Venipuncture; Near Infrared Light; Paediatric venepuncture; Venous blood sampling
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Venipuncture without near-infrared light
- Experimental group (Experimental): Venipuncture with near-infrared light
  Interventions: Procedure: venipuncture with near-infrared light

INTERVENTIONS:
Procedure: venipuncture with near-infrared light — with near-infrared light to locate the veins
  Arms: Experimental group

SUMMARY:
The purpose of this study is to determine whether the act of venipuncture is more successful on the first attempt using near infrared light compared to a standard puncture on children or newborn whose venous access is considered difficult due to lack of visibility of the veins.

DETAILED DESCRIPTION:
This trial aims to evaluate the act of venipuncture with or without the near-infrared light device for any children requiring a venipuncture for a blood sample or for insertion of peripheral venous line in neonatal intensive care and neonatology, and in pediatric emergencies.

For any eligible patient, at least one parent will be approached by a member of the medical or paramedical team trained on the protocol to explain the study to him/her and to be able to include the child during the next venous blood sampling or the insertion of a venous line. In case the parent agrees on the child's participation, the investigator is in charge of obtaining an informed consent.

During the next venous blood sampling or the insertion of a venous line, the nurse responsible for the patient:

* Takes the next consecutively numbered randomization envelope from the room intended for this purpose. This envelope is opaque and contains the randomization group in which the child is assigned (near infrared light or standard technique)
* Takes a study observation book located in the room intended for this purpose.
* Once the nurse is ready to do the venipuncture and before having identified the vein to be punctured, he/she opens the envelope to find out whether or not near infrared light will be used for spotting the vein to be punctured while the person (caregiver or nurse) who will help him during the procedure is present.
* Venous blood sampling or insertion of a venous line according to the technique indicated by the randomization (near infrared light or standard technique) for the first attempt at venipuncture.
* If the first venipuncture attempt fails, the nurse can chose to carry out the 2nd or 3rd attempt with or without near infrared light. Only the first 3 attempts progress will be recorded in the observation book.
* When the venous blood drawing or the insertion of a venous line is over, whether it is successful or not, the assistant present during the procedure completes the observation book on the sampling part.
* The notebook and the envelope used are stored in the room intended for this purpose.

To avoid device-related bias, the AccuVein® AV 400 (CE 0086 marking) was chosen. This device uses near infrared light to detect superficial veins under the skin and then projects an image of these veins onto the skin surface, exactly above the veins. The device will be held between 10 and 20 cm perpendicular to the skin, because at this distance the projected image corresponds to the actual size of the veins located below the skin. It will be either attached to an articulated arm in order to free the operator's hands to perform the procedure, or held by an assistant above the venipuncture site. The assistant can reorient the device during the procedure. The light from the AccuVein® device should not be aimed at the child's eyes. In neonatal intensive care and neonatology, during any use, the newborn's eyes will be covered during the procedure's implementation.

ELIGIBILITY:
Inclusion Criteria

* Any child aged at most 44 weeks + 6 days of corrected term hospitalized in neonatal intensive care and neonatology with a medical prescription for a venous blood sample or for insertion of a peripheral venous line and with visibility and palpability of the vein under 5mm

  *OR
* Any child under the age of 18 in the emergency room with a prescription for a blood test or for insertion of a peripheral venous line and with visibility and palpability of the vein under 5mm
* One parent agreed on their child participation in this study.
* Patient with health insurance

Exclusion Criteria

* Vital emergency which needs a venous route instalment
* Parental refusal
* Parents who do not speak French
* Patient who has already been included in the study
* Blood sample taken by a medical student or a nursing student or childcare nurse student.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
First venipuncture attempt | at day 0
  Obtention 0.5 ml of blood injection of 1.5 ml of physiological serum without extravasation after the first blood sampling attempt or the first attempt of a peripheral venous line.

SECONDARY OUTCOMES:
Successful venepuncture duration | at day 0
  Duration from application of tourniquet to obtention of 0.5 ml of blood After the first blood sampling attempt or the first attempt of a peripheral venous line at most after the 3rd venepuncture attempt
Pain evaluation during venipuncture | at day 0
  Using FLACC or DAN (acute pain of the new-born) scale (score 0 to 10, 10 is most painful) at most after the 3rd venepuncture attempt
Caregivers's opinion | at day 0
  Opinion of caregivers on the ease of use, effectiveness and their general satisfaction, using a small questionary (very unsatisfied, unsatisfied, satisfied, very satisfied) at most after the 3rd venepuncture attempt

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo CARBAJAL, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No